CLINICAL TRIAL: NCT06788067
Title: Impact of Time Interval Between Trauma and Operation on Clinical Outcome in Patients With Delayed Rib Fixation (Nonunion)
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-02144; kt25Lardinois
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Rib Fractures; Nonunion of Fracture
Keywords: Surgical stabilization of rib fractures (SSRF); Delayed SSRF; Nonunion SSRF
MeSH Terms: conditions — Rib Fractures; Fractures, Ununited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delayed SSRF: Patients who underwent surgery between 3 weeks and 3 months after trauma
- Nonunion SSRF: Patients who underwent surgery more than 3 months after trauma

SUMMARY:
The goal of this monocentric observational study is to evaluate the outcomes of patients who underwent a delayed surgical stabilization of rib fractures/surgical stabilization of rib fracture nonunion (SSRFN) based on the timing of surgery after trauma.

DETAILED DESCRIPTION:
Rib fractures occur in a significant number of patients with blunt chest trauma, and while conservative treatment remains the standard, surgical stabilization of rib fractures (SSRF) has shown improved clinical outcomes. However, conservative therapy often results in chronic chest pain and long-term incapacity, with up to 64% of patients experiencing persistent pain. Additionally, rib fracture nonunion, a condition where the bone fails to heal, affects approximately 12-15% of cases treated conservatively and can lead to long-term complications, including pain, limited mobility, and impaired quality of life.

This single-center observational study aims to analyze the outcomes of patients who underwent delayed SSRF (surgery between 3 weeks and 3 months after trauma) or nonunion SSRF (surgery performed more than 3 months after trauma). To assess whether a shorter interval between trauma and surgery results in better outcomes, the primary objective is to assess the persistence of thoracic pain in both patient groups. The secondary objective is to determine if SSRF improved patients' well-being.

This prospective research project is a single center analysis of existing data on patients, who underwent rib fixation for nonunion at the Department of Thoracic Surgery of the University Hospital Basel between January 1st, 2012 and June 30th, 2024. A prospective follow-up visit will be organized to assess the postoperative outcome.

The results of this study will provide valuable insights into optimizing treatment timelines for non consolidated rib fractures or rib fracture nonunion, improving patient outcomes and reducing long-term pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the study specific consent form
* Patients aged ≥18 years at the time of informed consent
* Patients who provided written informed consent in accordance with ICH-GCP regulations prior to participating any protocol-specific follow-up
* Patients with at least one rib fracture caused by trauma (traffic accident, falls), surgery (cardiac, thoracic, lung transplantation), sports, cough, and cardiopulmonary resuscitation

Exclusion Criteria:

* Patients who were treated conservatively
* Patients who underwent rib fixation till 3 weeks after trauma
* Patients who underwent SSRF prior to SSRFN
* Patients who are unable to follow the procedures of the study, e. g. have insufficient knowledge of German or French languages, psychological disorders, dementia etc.
* Patients with a pathological rib fracture(s) due to malignancy or radiation
* Participation in any interventional study in our department that might influence any of the outcome parameters
* Patients who underwent an initial surgery of rib fracture prior to development of a rib fracture nonunion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 75-80, patients who underwent rib fixation later than 3 weeks after trauma at the Department of Thoracic Surgery of the University Hospital Basel between 2012 and end of June 2024
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain status at Follow-up (FU) | After surgery at follow-up visit (1-8 weeks after recruitment)
  The pain status at the timepoint of the follow-up visit is measured using the numeric rating scale (NRS, scale 0: no pain to 10: worst pain) in different situations (at rest, at movement, and during deep inspiration). The type of pain (local, diffuse, neurogenic) will be also assessed.
Recommendation of the surgery to another person in a situation like the own | After surgery at follow-up visit (1-8 weeks after recruitment)
  The patients will be asked if they would recommend the surgery to another person in a situation like the own. The assessment will be performed in two categories: yes/no.
Pain status at FU compared to before surgery | After surgery at follow-up visit (1-8 weeks after recruitment)
  The pain status at the timepoint of the follow-up visit compared to the timepoint before surgery in five distinct categories on a Likert-scale (much better, slightly better, no change, slightly worse, much worse).
Painkiller Use (including nonsteroidal anti-inflammatory drugs and opioids) | After surgery at follow-up visit (1-8 weeks after recruitment)
  The painkiller use including nonsteroidal anti-inflammatory drugs and opioids is being recorded.

SECONDARY OUTCOMES:
Health status | After surgery at follow-up visit (1-8 weeks after recruitment)
  The subjective health-related quality of life is recorded using the 12-Item Short-Form (SF-12) questionnaire. The SF-12 is a validated scale used to assess physical and mental health, with scores ranging from 0 to 100, where higher scores indicate better health and well-being.
Resumption of daily/professional activity at FU | After surgery at follow-up visit (1-8 weeks after recruitment)
  Resumption of former professional activity and daily activities will be assessed by use of the numeric rating scale (NRS, scale 0: no pain to 10: worst pain).
Resumption of daily/professional activity at FU compared to before surgery | After surgery at follow-up visit (1-8 weeks after recruitment)
  Resumption of former professional activity and daily activities will be assessed by comparison with the situation before trauma and before surgery (much better, slightly better, no change, slightly worse, much worse).
Complications | Day 30 after surgery
  Complications related to surgery until/at 30 d after surgery according to the Clavien-Dindo classification.
Correlation between Number of Broken Ribs, Fixed Ribs, and Impact on Patient Outcomes | After surgery at follow-up visit (1-8 weeks after recruitment)
  This outcome assesses the relationship between the number of broken ribs, the number of surgically fixed ribs, and their influence on patient recovery and clinical outcomes.
Association between Age and clinical outcomes | After surgery at follow-up visit (1-8 weeks after recruitment)
  This outcome measures the association between patient age and the clinical outcomes following rib fractures.
Impact of Gender and Clinical Outcomes | After surgery at follow-up visit (1-8 weeks after recruitment)
  This outcome measures the impact of patient's gender and clinical outcomes following rib fractures
Impact of Rib Fracture Localization on Clinical Outcomes | After surgery at follow-up visit (1-8 weeks after recruitment)
  This outcome measures the impact of the location of rib fractures on clinical outcomes.
Frequency of Risk Factors for Rib Fracture Nonunion | After surgery at follow-up visit (1-8 weeks after recruitment)
  Frequency of risk factors for nonunion like nicotine use, diabetes mellitus, medication use including nonsteroidal anti-inflammatory drugs and opioids, osteoporosis, hypothyroidism.
Physical examination | After surgery at follow-up visit (1-8 weeks after recruitment)
  The incidence of chest wall instability and persistent clicking is assessed at the FU visit by a physical examination.

OTHER OUTCOMES:
Satisfaction with the decision for surgery | After surgery at follow-up visit (1-8 weeks after recruitment)
  Satisfaction with the decision for surgery will be assessed by use of NRS (numerical rating scale). (Would you have let the surgery done again? 0=Yes, absolutely satisfied; 10= absolutely dissatisfied):
Satisfaction with cosmetic results | After surgery at follow-up visit (1-8 weeks after recruitment)
  Satisfaction with cosmetic results of the surgery will be assessed with numeric rating scale (NRS: 0= absolutely satisfied; 10= absolutely dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Svec, Principal Investigator — Department of Thoracic Surgery, University Hospital Basel
Locations (1):
- Department of Thoracic Surgery, University Hospital Basel, Basel, Canton of Basel-City, Switzerland